CLINICAL TRIAL: NCT01221558
Title: Effects of Lycopene Supplementation on Oxidative Stress and Markers of Endothelial Function in Healthy Men
Brief Title: Effects of Lycopene on Oxidative Stress and Markers of Endothelial Function Healthy Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: principal investigator : Jong Ho Lee, Ph.D., Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: L-01
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Men
MeSH Terms: interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6mg lycopene (Experimental)
  Interventions: Dietary Supplement: lycopene
- 15mg lycopene (Experimental)
  Interventions: Dietary Supplement: lycopene
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: lycopene

INTERVENTIONS:
Dietary Supplement: lycopene

SUMMARY:
The hypothesis was that an increase in serum lycopene levels following supplementation with capsules containing natural lycopene rich tomato extract would reduce oxidative stress and improve endothelial function in healthy men with low intake of fruits and vegetables. A randomized double-blind, placebo-controlled study was designed to assess the changes in serum lycopene levels, oxidative stress and endothelial function in response to an 8-week treatment with lycopene supplementation.

DETAILED DESCRIPTION:
The healthy men aged 20-60 years, who frequently smoked cigarettes or consumed alcohol, were enrolled in this study. Subjects were excluded if they consumed more than 3 servings/day of vegetables and fruit, or more than one serving/week of lycopene-rich foods; took antioxidant, vitamin, or mineral supplements; had any history of chronic disease; or were taking lipid-lowering or antihypertensive medications.The subjects were randomly assigned to receive placebo, 6mg, or 15mg lycopene capsule per day for 8 weeks. Study substances were suspended in soybean oil and given in acid-soluble gelatin capsules. A placebo containing soybean oil (100%) was supplied in identical-looking capsules. All the subjects were instructed to consume one capsule per day right after any meal of their choice. All participants were encouraged to maintain their usual lifestyle and dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* healthy men who frequently smoked cigarettes or consumed alcohol

Exclusion Criteria:

* consumption of more than 3 servings/day of vegetables and fruit, or more than one serving/week of lycopene-rich foods
* taking antioxidant, vitamin, or mineral supplements
* any history of chronic disease (diabetes, heart disease, renal disease)
* taking lipid-lowering or antihypertensive medications

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
lymphocyte DNA damage | 8 weeks
antioxidant enzymes : SOD, GSH-Px, Catalase | 8 weeks
lipid peroxidation marker : MDA, urinary 8 epi-PGF 2alpha | 8 weeks
oxidized LDL | 8 weeks

SECONDARY OUTCOMES:
Reactive hyperemia peripheral arterial tonometry (RH-PAT) index | 8 weeks
VCAM-1/ICAM-1 | 8 weeks
cytokines : IL-6, TNF-alpha, IL-1beta | 8 weeks
hs-CRP | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea